CLINICAL TRIAL: NCT06763653
Title: A Prospective, Multi-Center, Randomized, Controlled Trial to Compare the Safety and Efficacy of Ultra Low Frequency Spinal Cord Stimulation Plus Conservative Medical Management (CMM) to CMM Alone in the Treatment of Chronic Axial Low Back Pain With Prominent Nociceptive Etiology - The FULFILL Study
Brief Title: Ultra Low Frequency Neuromodulation for Nociceptive Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Presidio Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMH-006
Record Dates: First submitted 2025-01-01; First posted 2025-01-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Nociceptive Pain; Axial Back Pain
Keywords: Neuromodulation; Spinal cord stimulation; Chronic low back pain
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Intervention Model Description: Option to crossover to alternate treatment arm at 6 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ULF therapy plus CMM (Experimental): An implanted SCS device delivering ultra low frequency neuromodulation
  Interventions: Device: ULF therapy; Other: CMM
- CMM alone (Active Comparator): Conventional medical management
  Interventions: Other: CMM

INTERVENTIONS:
Device: ULF therapy — ultra low frequency spinal cord stimulation
  Arms: ULF therapy plus CMM
Other: CMM — conventional medical management

SUMMARY:
The goal of this clinical trial is to learn if Ultra Low Frequency (ULF) neuromodulation works to treat nociceptive chronic low back pain in adults. It will also evaluate the safety of ULF therapy. The main questions it aims to answer are:

* Does ULF neuromodulation reduce chronic low back pain?
* What, if any, unexpected medical problems do participants experience when treated with ULF neuromodulation?

Researchers will compare ULF therapy to conventional treatments for chronic low back pain. Participants will:

* Be randomly assigned to either the study device or to conventional medical treatments
* Undergo standard surgical procedures to place the study device if assigned to the device arm
* Attend regular clinic visits over 24 months for checkups and data collection

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, controlled trial in which subjects with chronic, intractable axial low back pain with prominent nociceptive features will be randomized 2:1 into either Ultra Low Frequency (ULF) therapy combined with conventional medical management (CMM) or CMM alone. The purpose of this study is to compare the safety and efficacy of ULF neuromodulation to CMM in Subjects with chronic, intractable axial low back pain with prominent nociceptive features over a 24-month period.

Subjects assigned to CMM will continue with further optimization of the best available medical treatments. Subjects assigned to ULF therapy will proceed with a temporary trial phase and be eligible for permanent device implant if they experience at least 50% back pain relief. An option to cross over to the alternative treatment arm will be permitted at the 6-month timepoint for subjects who meet the criteria. The study primary endpoint will be evaluated at 3 months and follow-up will continue for 24 months total.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic, intractable nociceptive axial low back pain with or without leg pain (VAS ≥6 cm for back pain over 7 days) for a minimum of 3 months.
2. Symptoms have failed to respond adequately to conservative therapies, including: physical therapy/exercise, medications, and interventional therapies.
3. Back pain greater than leg pain.
4. ODI score ≥30 and ≤80.
5. On stable pain medications or on no pain medications.
6. Considered medically stable and a suitable surgical candidate.
7. Able to operate the device.
8. Willing to sign the Human Research Ethics Committee (HREC)/Institutional Review Board (IRB) approved informed consent form.
9. Willing and deemed capable of complying with the requirements of the study protocol, including attending all scheduled visits.
10. Twenty-two (22) years of age or older.
11. Able to complete questionnaires independently.

Exclusion Criteria:

1. Have a systemic condition or disease not stabilized or judged by the investigator to be incompatible with participation in the study.
2. Suffer from severe cognitive impairment that would impair ability to complete subject questionnaires or operation of the device.
3. Diagnosed with an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance, intervention and/or ability to evaluate treatment outcome as assessed by a clinical psychologist or psychiatrist.
4. Presence of spinal stenosis, structural spinal abnormality, or spinal instrumentation observed on MRI or CT that would make lead placement unsafe or untowardly difficult.
5. Previous experience with neuromodulation devices for pain.
6. Opioid usage with average total daily morphine equivalent dose (MED) of >100 mg.
7. Have an untreated addiction to alcohol or other drugs within 6 months of screening visit.
8. Have a cardiac demand pacemaker, implanted defibrillator, or another implanted electronic device.
9. Have a known hypersensitivity to any of the procedural agents or materials in the study device that is inserted into the subject.
10. Have a known need for an MRI or surgery through the end of the study.
11. Candidates of child-bearing potential cannot be pregnant nor plan to become pregnant during the study.
12. Diagnosed with untreated malicious or malignant neoplasms or have a life expectancy of less than 1 year.
13. Be participating in another interventional clinical trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Back pain VAS responder rate at 3 months | 3 months
  Comparison between the groups of the proportion of participants achieving at least 50% back pain relief from baseline, measured on a 10 cm visual analog scale (VAS).

SECONDARY OUTCOMES:
Composite of back pain relief measured by VAS and functional improvement measured by ODI at 6 months | 6 months
  Comparison between the groups of the proportion of participants who are both back pain responders (at least 50% relief from baseline VAS) and have at least a 10 point improvement in disability from baseline as measured by Oswestry Disability Index (ODI).
Back pain VAS responder rate at 6 months | 6 months
  Comparison between the groups of the proportion of participants achieving at least 50% back pain relief from baseline, measured on a 10 cm visual analog scale (VAS).
Functional improvement measured by ODI at 6 months | 6 months
  Comparison between the groups of the proportion of participants who have at least a 10 point improvement in disability from baseline as measured by Oswestry Disability Index (ODI).
Average change in back pain VAS at 3 months | 3 months
  Comparison between the groups in the average percentage change from baseline in back pain intensity, measured on a 10 cm visual analog scale (VAS).
Average change in back pain VAS at 6 months | 6 months
  Comparison between the groups in the average percentage change from baseline in back pain intensity, measured on a 10 cm visual analog scale (VAS).
Average change in disability measured by ODI at 3 months | 3 months
  Comparison between the groups in the average change from baseline in disability, measured by the Oswestry Disability Index (ODI).
Average change in disability measured by ODI at 6 months | 6 months
  Comparison between the groups in the average change from baseline in disability, measured by the Oswestry Disability Index (ODI).
Average change in health-related quality of life assessed by EQ-5D-5L at 6 months | 6 months
  Comparison between the groups in the average change from baseline in health-related quality of life, measured by the EuroQol Index (EQ-5D-5L).
Back pain VAS remitter rate at 6 months | 6 months
  Comparison between the groups of the proportion of participants achieving back pain remission from baseline, defined as a score of 3 cm or less for 6 consecutive months, measured on a 10 cm visual analog scale (VAS).
Leg pain VAS responder rate at 3 months | 3 months
  Among subjects with baseline leg pain VAS of at least 5 cm, comparison between the groups of the proportion of participants achieving at least 50% leg pain relief from baseline, measured on a 10 cm visual analog scale (VAS).
Leg pain VAS responder rate at 6 months | 6 months
  Among subjects with baseline leg pain VAS of at least 5 cm, comparison between the groups of the proportion of participants achieving at least 50% leg pain relief from baseline, measured on a 10 cm visual analog scale (VAS).
Average change in opioid dose at 6 months | 6 months
  Comparison between the groups in the average change from baseline in opioid equivalent medication dosage.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - The International Spine Centre, Norwood, South Australia
  - CerCare Pty Ltd, Wayville, South Australia
  - Monash House Research Centre, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No